CLINICAL TRIAL: NCT02373930
Title: A Phase I, 2-part Relative Oral Bioavailability Study of Different Fixed Dose Combinations of Dolutegravir and Rilpivirine in Fasted and Fed Healthy Subjects
Brief Title: Relative Oral Bioavailability Study of Different Fixed Dose Combinations of Dolutegravir and Rilpivirine in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Janssen Pharmaceuticals (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 201674
Record Dates: First submitted 2015-02-23; First posted 2015-02-27 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-06

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: Dolutegravir; safety; Rilpivirine; fixed dose combination; relative bioavailability
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — dolutegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (15):
- Part 1 Cohort 1- Sequence 1 (Experimental): Each subject will receive a single dose of Treatment A (DTG 50 mg tablet plus RPV 25 mg tablet), Treatment B (DTG/RPV 50 mg/25 mg: Product Code AS) and Treatment C (DTG/RPV 50 mg/25 mg: Product Code AM) in period 1, period 2 and period 3 respectively with a washout period of >=9 days between doses of study medication. All treatments will be administered in fed state.
  Interventions: Drug: DTG 50 mg; Drug: RPV 25 mg; Drug: DTG/RPV 50 mg/25 mg: Product Code AS; Drug: DTG/RPV 50 mg/25 mg: Product Code AM
- Part 1 Cohort 1- Sequence 2 (Experimental): Each subject will receive a single dose of Treatment D (DTG/RPV 50 mg/25 mg: Product Code AQ), Treatment A (DTG 50 mg tablet plus RPV 25 mg tablet) and Treatment B (DTG/RPV 50 mg/25 mg: Product Code AS) in period 1, period 2 and period 3 respectively with a washout period of >=9 days between doses of study medication. All treatments will be administered in fed state.
  Interventions: Drug: DTG 50 mg; Drug: RPV 25 mg; Drug: DTG/RPV 50 mg/25 mg: Product Code AS; Drug: DTG/RPV 50 mg/25 mg: Product Code AQ
- Part 1 Cohort 1- Sequence 3 (Experimental): Each subject will receive a single dose of Treatment B (DTG/RPV 50 mg/25 mg: Product Code AS), Treatment E (DTG/RPV 50 mg/25 mg: Product Code AK) and Treatment A (DTG 50 mg tablet plus RPV 25 mg tablet) in period 1, period 2 and period 3 respectively with a washout period of >=9 days between doses of study medication. All treatments will be administered in fed state.
  Interventions: Drug: DTG 50 mg; Drug: RPV 25 mg; Drug: DTG/RPV 50 mg/25 mg: Product Code AS; Drug: DTG/RPV 50 mg/25 mg: Product Code AK
- Part 1 Cohort 1- Sequence 4 (Experimental): Each subject will receive a single dose of Treatment A (DTG 50 mg tablet plus RPV 25 mg tablet), Treatment C (DTG/RPV 50 mg/25 mg: Product Code AM) and Treatment D (DTG/RPV 50 mg/25 mg: Product Code AQ) in period 1, period 2 and period 3 respectively with a washout period of >=9 days between doses of study medication. All treatments will be administered in fed state.
  Interventions: Drug: DTG 50 mg; Drug: RPV 25 mg; Drug: DTG/RPV 50 mg/25 mg: Product Code AM; Drug: DTG/RPV 50 mg/25 mg: Product Code AQ
- Part 1 Cohort 1- Sequence 5 (Experimental): Each subject will receive a single dose of Treatment C (DTG/RPV 50 mg/25 mg: Product Code AM), Treatment A (DTG 50 mg tablet plus RPV 25 mg tablet), and Treatment E (DTG/RPV 50 mg/25 mg: Product Code AK) in period 1, period 2 and period 3 respectively with a washout period of >=9 days between doses of study medication. All treatments will be administered in fed state.
  Interventions: Drug: DTG 50 mg; Drug: RPV 25 mg; Drug: DTG/RPV 50 mg/25 mg: Product Code AM; Drug: DTG/RPV 50 mg/25 mg: Product Code AK
- Part 1 Cohort 1- Sequence 6 (Experimental): Each subject will receive a single dose of Treatment E (DTG/RPV 50 mg/25 mg: Product Code AK), Treatment D (DTG/RPV 50 mg/25 mg: Product Code AQ) and Treatment A (DTG 50 mg tablet plus RPV 25 mg tablet), in period 1, period 2 and period 3 respectively with a washout period of >=9 days between doses of study medication. All treatments will be administered in fed state.
  Interventions: Drug: DTG 50 mg; Drug: RPV 25 mg; Drug: DTG/RPV 50 mg/25 mg: Product Code AQ; Drug: DTG/RPV 50 mg/25 mg: Product Code AK
- Part 2 Cohort 2- Sequence 1 (Experimental): Each subject will receive a single dose of Treatment F (DTG/RPV FDC-1) in fasted state, Treatment F (DTG/RPV FDC-1) in fed state and Treatment A (DTG 50 mg tablet plus RPV 25 mg tablet) in fasted state in period 1, period 2 and period 3 respectively with a washout period of >=9 days between doses of study medication.
  Interventions: Drug: DTG 50 mg; Drug: RPV 25 mg; Drug: DTG/RPV 50 mg/25 mg: Product Code AS; Drug: DTG/RPV 50 mg/25 mg: Product Code AM; Drug: DTG/RPV 50 mg/25 mg: Product Code AQ; Drug: DTG/RPV 50 mg/25 mg: Product Code AK; Drug: DTG/RPV 50 mg/25 mg: Product Code AR
- Part 2 Cohort 2- Sequence 2 (Experimental): Each subject will receive a single dose of Treatment F (DTG/RPV FDC-1) in fed state, Treatment A (DTG 50 mg tablet plus RPV 25 mg tablet) in fasted state and Treatment F (DTG/RPV FDC-1) in fasted state in period 1, period 2 and period 3 respectively with a washout period of >=9 days between doses of study medication.
  Interventions: Drug: DTG 50 mg; Drug: RPV 25 mg; Drug: DTG/RPV 50 mg/25 mg: Product Code AS; Drug: DTG/RPV 50 mg/25 mg: Product Code AM; Drug: DTG/RPV 50 mg/25 mg: Product Code AQ; Drug: DTG/RPV 50 mg/25 mg: Product Code AK; Drug: DTG/RPV 50 mg/25 mg: Product Code AR
- Part 2 Cohort 2- Sequence 3 (Experimental): Each subject will receive a single dose of Treatment A (DTG 50 mg tablet plus RPV 25 mg tablet) in fasted state, Treatment F (DTG/RPV FDC-1) in fasted state and Treatment F (DTG/RPV FDC-1) in fed state in period 1, period 2 and period 3 respectively with a washout period of >=9 days between doses of study medication.
  Interventions: Drug: DTG 50 mg; Drug: RPV 25 mg; Drug: DTG/RPV 50 mg/25 mg: Product Code AS; Drug: DTG/RPV 50 mg/25 mg: Product Code AM; Drug: DTG/RPV 50 mg/25 mg: Product Code AQ; Drug: DTG/RPV 50 mg/25 mg: Product Code AK; Drug: DTG/RPV 50 mg/25 mg: Product Code AR
- Part 2 Cohort 3- Sequence 4 (Experimental): Each subject will receive a single dose of Treatment G (DTG/RPV FDC-2) in fasted state, Treatment G (DTG/RPV FDC-2) in fed state and Treatment A (DTG 50 mg tablet plus RPV 25 mg tablet) in fasted state in period 1, period 2 and period 3 respectively with a washout period of >=9 days between doses of study medication.
  Interventions: Drug: DTG 50 mg; Drug: RPV 25 mg; Drug: DTG/RPV 50 mg/25 mg: Product Code AS; Drug: DTG/RPV 50 mg/25 mg: Product Code AM; Drug: DTG/RPV 50 mg/25 mg: Product Code AQ; Drug: DTG/RPV 50 mg/25 mg: Product Code AK; Drug: DTG/RPV 50 mg/25 mg: Product Code AR
- Part 2 Cohort 3- Sequence 5 (Experimental): Each subject will receive a single dose of Treatment G (DTG/RPV FDC-2) in fed state, Treatment A (DTG 50 mg tablet plus RPV 25 mg tablet) in fasted state and Treatment G (DTG/RPV FDC-2) in fasted state in period 1, period 2 and period 3 respectively with a washout period of >=9 days between doses of study medication.
  Interventions: Drug: DTG 50 mg; Drug: RPV 25 mg; Drug: DTG/RPV 50 mg/25 mg: Product Code AS; Drug: DTG/RPV 50 mg/25 mg: Product Code AM; Drug: DTG/RPV 50 mg/25 mg: Product Code AQ; Drug: DTG/RPV 50 mg/25 mg: Product Code AK; Drug: DTG/RPV 50 mg/25 mg: Product Code AR
- Part 2 Cohort 3- Sequence 6 (Experimental): Each subject will receive a single dose of Treatment A (DTG 50 mg tablet plus RPV 25 mg tablet) in fasted state and Treatment G (DTG/RPV FDC-2) fasted state and Treatment G (DTG/RPV FDC-2) in fed state in period 1, period 2 and period 3 respectively with a washout period of >=9 days between doses of study medication.
  Interventions: Drug: DTG 50 mg; Drug: RPV 25 mg; Drug: DTG/RPV 50 mg/25 mg: Product Code AS; Drug: DTG/RPV 50 mg/25 mg: Product Code AM; Drug: DTG/RPV 50 mg/25 mg: Product Code AQ; Drug: DTG/RPV 50 mg/25 mg: Product Code AK; Drug: DTG/RPV 50 mg/25 mg: Product Code AR
- Part 2 Cohort 4- Sequence 7 (Experimental): Each subject will receive a single dose of Treatment H (DTG/RPV FDC-3) in fasted state, Treatment H (DTG/RPV FDC-3) in fed state and Treatment A (DTG 50 mg tablet plus RPV 25 mg tablet) in fasted state in period 1, period 2 and period 3 respectively with a washout period of >=9 days between doses of study medication.
  Interventions: Drug: DTG 50 mg; Drug: RPV 25 mg; Drug: DTG/RPV 50 mg/25 mg: Product Code AS; Drug: DTG/RPV 50 mg/25 mg: Product Code AM; Drug: DTG/RPV 50 mg/25 mg: Product Code AQ; Drug: DTG/RPV 50 mg/25 mg: Product Code AK; Drug: DTG/RPV 50 mg/25 mg: Product Code AR
- Part 2 Cohort 4- Sequence 8 (Experimental): Each subject will receive a single dose of Treatment H (DTG/RPV FDC-3) in fed state, Treatment A (DTG 50 mg tablet plus RPV 25 mg tablet) in fasted state and Treatment H (DTG/RPV FDC-3) in fasted state in period 1, period 2 and period 3 respectively with a washout period of >=9 days between doses of study medication.
  Interventions: Drug: DTG 50 mg; Drug: RPV 25 mg; Drug: DTG/RPV 50 mg/25 mg: Product Code AS; Drug: DTG/RPV 50 mg/25 mg: Product Code AM; Drug: DTG/RPV 50 mg/25 mg: Product Code AQ; Drug: DTG/RPV 50 mg/25 mg: Product Code AK; Drug: DTG/RPV 50 mg/25 mg: Product Code AR
- Part 2 Cohort 4- Sequence 9 (Experimental): Each subject will receive a single dose of Treatment A (DTG 50 mg tablet plus RPV 25 mg tablet) in fasted state and Treatment H (DTG/RPV FDC-3) fasted state and Treatment H (DTG/RPV FDC-3) in fed state in period 1, period 2 and period 3 respectively with a washout period of >=9 days between doses of study medication.
  Interventions: Drug: DTG 50 mg; Drug: RPV 25 mg; Drug: DTG/RPV 50 mg/25 mg: Product Code AS; Drug: DTG/RPV 50 mg/25 mg: Product Code AM; Drug: DTG/RPV 50 mg/25 mg: Product Code AQ; Drug: DTG/RPV 50 mg/25 mg: Product Code AK; Drug: DTG/RPV 50 mg/25 mg: Product Code AR

INTERVENTIONS:
Drug: DTG 50 mg — Dolutegravir will be supplied as a white, film-coated, round tablet with a unit dose strength of 50 mg to be administered orally
Drug: RPV 25 mg — Rilpivirine will be supplied as a white to off-white, film-coated, round biconvex tablet with a unit dose strength of 25 mg to be administered orally
Drug: DTG/RPV 50 mg/25 mg: Product Code AS — DTG/RPV will be supplied as a pink, film coated, round biconvex tablet with a unit dose strength of 50 mg DTG and 25 mg RPV to be administered orally
  Arms: Part 1 Cohort 1- Sequence 1; Part 1 Cohort 1- Sequence 2; Part 1 Cohort 1- Sequence 3; Part 2 Cohort 2- Sequence 1; Part 2 Cohort 2- Sequence 2; Part 2 Cohort 2- Sequence 3; Part 2 Cohort 3- Sequence 4; Part 2 Cohort 3- Sequence 5; Part 2 Cohort 3- Sequence 6; Part 2 Cohort 4- Sequence 7; Part 2 Cohort 4- Sequence 8; Part 2 Cohort 4- Sequence 9
Drug: DTG/RPV 50 mg/25 mg: Product Code AM — DTG/RPV will be supplied as a pink, film coated, oval, biconvex tablet with a unit dose strength of 50 mg DTG and 25 mg RPV to be administered orally
  Arms: Part 1 Cohort 1- Sequence 1; Part 1 Cohort 1- Sequence 4; Part 1 Cohort 1- Sequence 5; Part 2 Cohort 2- Sequence 1; Part 2 Cohort 2- Sequence 2; Part 2 Cohort 2- Sequence 3; Part 2 Cohort 3- Sequence 4; Part 2 Cohort 3- Sequence 5; Part 2 Cohort 3- Sequence 6; Part 2 Cohort 4- Sequence 7; Part 2 Cohort 4- Sequence 8; Part 2 Cohort 4- Sequence 9
Drug: DTG/RPV 50 mg/25 mg: Product Code AQ — DTG/RPV will be supplied as a pink, film coated, round, biconvex tablet with a unit dose strength of 50 mg DTG and 25 mg RPV to be administered orally
  Arms: Part 1 Cohort 1- Sequence 2; Part 1 Cohort 1- Sequence 4; Part 1 Cohort 1- Sequence 6; Part 2 Cohort 2- Sequence 1; Part 2 Cohort 2- Sequence 2; Part 2 Cohort 2- Sequence 3; Part 2 Cohort 3- Sequence 4; Part 2 Cohort 3- Sequence 5; Part 2 Cohort 3- Sequence 6; Part 2 Cohort 4- Sequence 7; Part 2 Cohort 4- Sequence 8; Part 2 Cohort 4- Sequence 9
Drug: DTG/RPV 50 mg/25 mg: Product Code AK — DTG/RPV will be supplied as pink, film coated, oval, biconvex tablet with a unit dose strength of 50 mg DTG and 25 mg RPV to be administered orally
  Arms: Part 1 Cohort 1- Sequence 3; Part 1 Cohort 1- Sequence 5; Part 1 Cohort 1- Sequence 6; Part 2 Cohort 2- Sequence 1; Part 2 Cohort 2- Sequence 2; Part 2 Cohort 2- Sequence 3; Part 2 Cohort 3- Sequence 4; Part 2 Cohort 3- Sequence 5; Part 2 Cohort 3- Sequence 6; Part 2 Cohort 4- Sequence 7; Part 2 Cohort 4- Sequence 8; Part 2 Cohort 4- Sequence 9
Drug: DTG/RPV 50 mg/25 mg: Product Code AR — DTG/RPV will be supplied as a pink, film coated, round, biconvex tablet with a unit dose strength of 50 mg DTG and 25 mg RPV to be administered orally
  Arms: Part 2 Cohort 2- Sequence 1; Part 2 Cohort 2- Sequence 2; Part 2 Cohort 2- Sequence 3; Part 2 Cohort 3- Sequence 4; Part 2 Cohort 3- Sequence 5; Part 2 Cohort 3- Sequence 6; Part 2 Cohort 4- Sequence 7; Part 2 Cohort 4- Sequence 8; Part 2 Cohort 4- Sequence 9

SUMMARY:
Treatment of human immunodeficiency virus (HIV) infection requires daily oral administration of a combination of antiretroviral drugs to reduce the patient's HIV levels. Dolutegravir (DTG), a HIV-1 integrase inhibitor (INI), and Rilpivirine (RPV), a non-nucleoside HIV-1 reverse transcriptase inhibitor (NNRTI), are approved for the treatment of HIV infection. This study is aimed to evaluate the relative bioavailability and food effect of single doses of several experimental fixed dose combination (FDC) tablets of Dolutegravir 50 milligrams (mg) and Rilpivirine 25 mg (DTG/RPV 50 mg/25 mg) relative to co-administration of a single dose of the reference single entity products (DTG 50 mg and RPV 25 mg) in healthy adult subjects. This is a 2-part study. Part 1 will be conducted as a randomized, open label, 3-way, crossover design in 24 subjects. Part 1 will evaluate the relative bioavailability of up to 4 test formulations relative to the reference single entity products administered in fed state. Part 2 will be conducted as a randomized, open-label, 3-way crossover design in 3 distinct cohorts each with 12 subjects. Part 2 will evaluate the relative bioavailability of up to 3 most promising FDC formulation selected from Part 1 (DTG/RPV FDC-1, DTG/RPV FDC-2, DTG/RPV FDC-3) administered in fasted and fed state. Subjects will also receive the reference treatment from Part 1 co-administered under fasted conditions. This study will consist of a screening visit, three treatment periods each with a single dose of study drug separated by a washout of at least 9 days and a follow-up visit. The total duration of participation of a subject in this study will be approximately 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac evaluation (history, electrocardiogram [ECG]).
* A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator in consultation with the medical monitor if required agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >=50 kilograms (kg) (110 pounds [lbs]) for men and >=45 kg (99 lbs) for women and body mass index (BMI) within the range 18.5-31.0 kg/square meter (m^2) (inclusive).
* Male or Female- Female: Female subject of non-reproductive potential : is eligible to participate if she is not pregnant (as confirmed by a negative serum or urine human chorionic gonadotrophin [hCG] test), not lactating, and at least one of the following conditions applies: Pre-menopausal females with one of the following: documented tubal ligation, documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion, hysterectomy, documented bilateral oophorectomy.

Postmenopausal defined as 12 months of spontaneous amenorrhea; in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) and estradiol levels consistent with menopause (refer to laboratory reference ranges for confirmatory levels). Females on hormone replacement therapy (HRT) must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment.

Reproductive potential and agrees to follow one of the options listed below in the GlaxoSmithKline (GSK) modified list of highly effective methods for avoiding pregnancy in females of reproductive potential (FRP) requirements from 30 days prior to the first dose of study medication and until at least five terminal half-lives (10 days) after the last dose of study medication and completion of the follow-up visit.

GSK Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP)

This list does not apply to FRP with same sex partners, when this is their preferred and usual lifestyle or for subjects who are and will continue to be abstinent from penile-vaginal intercourse on a long term and persistent basis.

* Intrauterine device that meets the standard operating procedure (SOP) effectiveness criteria including a <1% rate of failure per year, as stated in the product label.
* Male partner sterilization with documentation of azoospermia prior to the female subject's entry into the study, and this male is the sole partner for that subject.
* Male condom combined with a vaginal spermicide (foam, gel, film, cream, or suppository).

These allowed methods of contraception are only effective when used consistently, correctly and in accordance with the product label. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.

Male:

* Male subjects with female partners of child bearing potential must comply with the following contraception requirements from the time of first dose of study medication until [at least five half-lives of study medication OR for a cycle of spermatogenesis following five terminal half-lives] after the last dose of study medication.

  1. Vasectomy with documentation of azoospermia.
  2. Male condom plus partner use of one of the contraceptive options below:
* Contraceptive subdermal implant that meets the SOP effectiveness criteria including a <1% rate of failure per year, as stated in the product label.
* Intrauterine device or intrauterine system that meets the SOP effectiveness criteria including a <1% rate of failure per year, as stated in the product label.
* Oral Contraceptive, either combined or progestrogen alone.
* Injectable progestrogen.
* Contraceptive vaginal ring.
* Percutaneous contraceptive patches.

These allowed methods of contraception are only effective when used consistently, correctly and in accordance with the product label. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.

* Capable of giving signed informed consent as described in protocol which includes compliance with the requirements and restrictions listed in the consent form and in this protocol.

Exclusion Criteria:

* Alanine aminotransferase (ALT) and bilirubin >1.5x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK medical monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 grams (g) of alcohol: 12 ounces (360 milliliter [mL]) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates their participation.
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment.
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* Where participation in the study would result in donation of blood or blood product in excess of 500 mL within 56 days.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Exclusion criteria for screening ECG (a single repeat is allowed for eligibility determination):

Heart Rate for males: <45 and >100 beats per minute (bpm), females: <50 and >100 bpm PR Interval for males: <120 and >220 milliseconds (msec) QRS Interval for males: <70 and >120 msec QT duration corrected for heart rate (QTc) interval (Fridericia's) for males: >450 msec Note: A heart rate from 100 to 110 bpm can be rechecked by ECG or vitals within 30 minutes to verify eligibility.

Evidence of previous myocardial infarction (does not include ST segment changes associated with repolarization).

Any conduction abnormality (including but not specific to left or right complete bundle branch block, atrioventricular block (AV block) (2nd degree or higher), Wolf Parkinson White [WPW] syndrome).

Sinus Pauses >3 seconds. Any significant arrhythmia which, in the opinion of the principal investigator OR GSK medical monitor, will interfere with the safety for the individual subject.

Non-sustained or sustained ventricular tachycardia (>=3 consecutive ventricular ectopic beats).

* Employment with Janssen and GSK or with the Investigator or study site, with direct involvement in the proposed study or other studies under the direction of that Investigator or study site, as well as family members of the employees or the Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2015-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Composite of pharmacokinetic (PK) parameters of a single dose of DTG and RPV administered together in a FDC tablet compared to co-administration of the single-entity DTG and RPV products in fed state (Part 1) | Part 1: Pre-dose and 0.25 hours (h), 0.5 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 4 h, 5 h, 6 h, 7 h, 9 h, 12 h, 16 h, 24 h, 48 h, 72 h, 120 h, and 168 hours post-dose in each treatment period.
  PK parameters will include area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUC [0-Infinity]), maximum observed concentration (Cmax) and apparent oral clearance (CL/F)
Composite of PK parameters of a single dose of DTG and RPV administered together in a FDC tablet compared to co-administration of the single-entity DTG and RPV products in fasted state (Part 2) | Part 2: Pre-dose and 0.25 h, 0.5 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 4 h, 5 h, 6 h, 7 h, 9 h, 12 h, 16 h, 24 h, 48 h, 72 h, 120 h, and 168 hours post-dose in each treatment period.
  PK parameters will include AUC (0-Infinity), Cmax and CL/F
Composite of PK parameters of DTG and RPV to evaluate the effect of food on the bioavailability of selected FDC formulation(s) of DTG and RPV (Part 2) | Part 2: Pre-dose and 0.25 h, 0.5 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 4 h, 5 h, 6 h, 7 h, 9 h, 12 h, 16 h, 24 h, 48 h, 72 h, 120 h, and 168 hours post-dose in each treatment period.
  PK parameters will include AUC (0-Infinity), Cmax and CL/F

SECONDARY OUTCOMES:
Composite of PK parameters of a single dose of DTG and RPV administered together in a FDC tablet compared to co-administration of the single-entity DTG and RPV products in fed state (Part 1) | Part 1: Pre-dose and 0.25 h, 0.5 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 4 h, 5 h, 6 h, 7 h, 9 h, 12 h, 16 h, 24 h, 48 h, 72 h, 120 h, and 168 hours post-dose in each treatment period.
  PK parameters will include area under the curve from time of dose administration to time of last quantifiable post-dose sample (AUC[0-t]), observed concentration at 24 h post-dose (C24), terminal elimination phase half-life (t1/2), lag time for absorption (tlag) and time to maximum observed concentration (tmax).
Composite of PK parameters of a single dose of DTG and RPV administered together in a FDC tablet compared to co-administration of the single-entity DTG and RPV products in fasted state (Part 2) | Part 2: Pre-dose and 0.25 h, 0.5 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 4 h, 5 h, 6 h, 7 h, 9 h, 12 h, 16 h, 24 h, 48 h, 72 h, 120 h, and 168 hours post-dose in each treatment period.
  PK parameters will include AUC (0-t), C24, t1/2, tlag and tmax.
Composite of PK parameters of DTG and RPV to evaluate the effect of food on the bioavailability of selected FDC formulation(s) of DTG and RPV (Part 2) | Part 2: Pre-dose and 0.25 h, 0.5 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 4 h, 5 h, 6 h, 7 h, 9 h, 12 h, 16 h, 24 h, 48 h, 72 h, 120 h, and 168 hours post-dose in each treatment period.
  PK parameters will include AUC (0-t), C24, t1/2, tlag and tmax.
Change from baseline in vital signs | Part 1 and 2: Baseline (Day 1) and up to Day 35
  Vital signs will include systolic and diastolic blood pressure and pulse rate
Number of subjects with adverse events (AEs) | Part 1 and 2: Up to Day 35
  AEs and serious adverse events (SAEs) will be collected from the start of study treatment until the follow-up contact.
Composite of clinical laboratory assessments | Part 1 and 2: Up to Day 35
  Clinical laboratory tests will include hematology, clinical chemistry, urinalysis parameters

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Overland Park, Kansas, United States